CLINICAL TRIAL: NCT03128996
Title: A Phase I/II Trial of Reduced Intensity Conditioning and Familial HLA-Mismatched Bone Marrow Transplantation in Children With Non-Malignant Disorders
Brief Title: Reduced Intensity Conditioning and Familial HLA-Mismatched BMT for Non-Malignant Disorders
Acronym: FAM BMT
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201611172
Record Dates: First submitted 2017-04-03; First posted 2017-04-26 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Severe Sickle Cell Disease; Bone Marrow Failure Syndromes; Metabolic Disorders; Immunologic Disorders; Hemoglobinopathies; Non-malignant Disorders
Keywords: Bone marrow transplant; Transplant; Transplantation; Reduced Intensity; Familial HLA mismatched
MeSH Terms: conditions — Anemia, Sickle Cell; Bone Marrow Failure Disorders; Metabolic Diseases; Immune System Diseases; Hemoglobinopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RIC Prep Regimen & GVHD Prophylaxis (Experimental): Single arm study. All patients receive the same Reduced Intensity Conditioning (RIC) regimen and GVHD prophylaxis regimen
  Interventions: Drug: RIC regimen; Drug: GVHD prophylaxis regimen

INTERVENTIONS:
Drug: RIC regimen — Days -60 to -21: hydroxyurea (30mg/kg/day po) >6hrs prior to 1st dose: alemtuzumab (3mg IV) Day -21: alemtuzumab (10mg IV or S/C) Day -20: alemtuzumab (15mg IV or S/C) (10mg if < 10kg) Day -19: alemtuzumab (20mg IV or S/C) (10mg if < 10kg) Days -8 to -4: fludarabine (30mg/m2/day IV) Day -4: thiotepa (8mg/kg IV) Day -3: melphalan (140mg/m2) Days -2 to -1: rest days/no therapy Day 0: bone marrow transplant
  Other Names: Transplant Preparative Regimen; Transplant Conditioning Regimen
Drug: GVHD prophylaxis regimen — Day +3 to +4: cyclophosphamide (50mg/kg/day IV) Day +5: Start of tacrolimus & Start of mycophenolate mofetil (MMF) Days +5, +14, +30, +60, +90: abatacept (IND) (10mg/kg/day IV) Day +90: rituximab (375mg/m2 IV once) Patients >/= 12 yrs - Days +120 to +180: abatacept (IND) monthly (10mg/kg/day IV) Patients >/= 12 yrs - Days +210 to +390: abatacept (IND) monthly (5mg/kg/day) Patients <12 yrs - Days +120 to +390: abatacept (IND) monthly (5mg/kg/day IV)
  Other Names: Graft versus Host Disease prophylaxis regimen

SUMMARY:
This study is designed to estimate the efficacy and toxicity of familial HLA mismatched bone marrow transplants in patients with non-malignant disease who are less than 21 years of age and could benefit from the procedure.

DETAILED DESCRIPTION:
Patients < 21 years of age with a non-malignant disorder benefited by hematopoietic stem cell transplant will receive a reduced intensity conditioning regimen consisting of hydroxyurea, alemtuzumab, fludarabine, thiotepa, and melphalan.

This will be followed by a familial HLA-mismatched bone marrow transplant. The primary objective is to establish safety and donor cell engraftment at 100 days and 1 year post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* Nonmalignant disorder requiring bone marrow transplant including bone marrow failure syndromes, metabolic disorders, immunologic disorders, or hemoglobinopathy
* For patients with sickle cell disease, must have one of the following severe manifestations:

  1. Overt or silent stroke or persistently elevated transcranial doppler velocities despite transfusion therapy
  2. Recurrent acute chest syndrome with significant respiratory compromise each time
  3. Sickle nephropathy
  4. Recurrent admissions for vaso-occlusive episodes resulting in prolonged opioid use and poor quality of life with interrupted school attendance activity
  5. Red cell alloimmunization with the need for chronic transfusions
  6. Recurrent osteonecrosis or multiple joint involvement from avascular necrosis
* Patients with sickle cell disease must have hemoglobin S < 30% within 30 days prior to beginning alemtuzumab
* Age </= 20.99 years at the time of enrollment
* Performance score >/= 50
* Left ventricular ejection fraction > 40% or left ventricular shortening fraction > 26% by echocardiogram
* DLCO > 40% (corrected for hemoglobin) or pulse oximetry with a baseline O2 saturation of >/= 90% on room air if too young to perform PFTs
* Serum creatinine </= 1.5x upper limit of normal for age and/or GFR > 70 mL/min/1.73m2
* Direct bilirubin < 2x upper limit of normal for age
* ALT and AST < 5x upper limit of normal for age
* Participants who have or are receiving >/= 8 packed red blood cell transfusions for >/= 1 year or >/= 20 packed red blood cell transfusions (lifetime cumulative) will undergo liver MRI for estimation of hepatic iron content.

  1. Liver biopsy is indicated for hepatic iron content >/= 7mg Fe/mg liver dry weight by liver MRI. Histologic examination of the liver must document for the absence of cirrhosis, bridging fibrosis, and active hepatitis
* Female subjects of childbearing potential, must agree to practice 2 methods of contraception at the same time from the time of signing of informed consent through 12 months post transplant. Male subjects must agree to practice effective barrier contraception or practice true abstinence from the time of signing informed consent through 12 months post transplant.
* Written informed consent must be obtained from all recipients in accordance with the guidelines of the institution's Human Studies Committee.

Exclusion Criteria:

* Patients who have an HLA-identical sibling who is able and willing to donate bone marrow
* Patients with cirrhosis or established bridging fibrosis of the liver or active hepatitis
* Uncontrolled bacterial, viral, or fungal infection within 6 weeks prior to enrollment
* Evidence of HIV infection or known HIV positive serology
* Patients who have received a previous stem cell transplant
* Patients who have received an investigational drug or device or off-label use of a drug or device within 3 months of enrollment
* Females who are pregnant or breast feeding
* Patients with active autoimmune disease (e.g. sarcoidosis, lupus, scleroderma)

Ages: 1 Day to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Estimated)
Dates: Start 2017-03-20 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2033-04 (Estimated)

PRIMARY OUTCOMES:
Donor engraftment | 100 days and 1 year post-transplant
  as measured by chimerism

SECONDARY OUTCOMES:
Time to neutrophil engraftment | 100 days post-transplant
  as measured by complete blood counts
Time to platelet engraftment | 100 days post-transplant
  as measured by complete blood counts
Effect of BMT on pulmonary function | 90 days, 1 year, and 2 years post-transplant
  as measured by pulmonary function tests
Effect of BMT on hepatic function | 90 days, 180 days, 1 year, and 2 years post-transplant
  as measured by laboratory evaluations
Effect of BMT on neurologic function | 90 days, 1 year, and 2 years post-transplant
  as measured by cognitive testing and quality of life surveys
Effect of BMT on cardiac function | 90 days, 1 year, and 2 years post-transplant
  as measured by echocardiograms
Effect of BMT on renal function | 90 days, 180 days, 1 year, and 2 years post-transplant
  as measured by laboratory evaluations
Pharmacokinetics of alemtuzumab | days -19, day 0, day +15, and day +30
  as measured by maximum plasma concentration of alemtuzumab
Pharmacokinetics of abatacept | days +30, +60, +90, 1 year, 1.5 years, and 2 years post-transplant
  as measured by maximum plasma concentration of abatacept
Incidence of acute graft-versus-host disease (GVHD) | 1 year post-transplant
  as measured by protocol grading scale
Incidence of chronic graft-versus-host disease (GVHD) | 2 years post-transplant
  as measured by protocol grading scale
Immune reconstitution | days +30, +60, +90, 1 year, 1.5 years, and 2 years post-transplant
  as measured by research laboratory evaluations

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Shenoy, MD, Principal Investigator — Washington University School of Medicine
Locations (4):
- United States (4):
  - Yale School of Medicine, New Haven, Connecticut
  - Nemours Children's Health, Wilmington, Delaware
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ngwube A, Shah N, Godder K, Jacobsohn D, Hulbert ML, Shenoy S. Abatacept is effective as GVHD prophylaxis in unrelated donor stem cell transplantation for children with severe sickle cell disease. Blood Adv. 2020 Aug 25;4(16):3894-3899. doi: 10.1182/bloodadvances.2020002236. PMID 32813873